CLINICAL TRIAL: NCT02538536
Title: A Phase 2, Open-label, Single Arm, Exploratory, Observational Study to Evaluate the Safety and Tolerability of PBI-4050 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Phase 2 Study to Evaluate the Safety and Tolerability of PBI-4050 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liminal BioSciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBI-4050-ATX-9-03
Record Dates: First submitted 2015-08-25; First posted 2015-09-02 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — setogepram

ARMS (1):
- PBI4050 (Experimental): Four 200 mg capsules (total 800 mg) administered orally, once daily.
  Interventions: Drug: PBI4050

INTERVENTIONS:
Drug: PBI4050

SUMMARY:
This is a Phase 2, open-label, single-arm study of the safety and tolerability of PBI-4050 800 mg daily oral administration in 40 adult patients with IPF.

DETAILED DESCRIPTION:
This Phase 2 multi-centre study will be performed by 6 Canadian sites. It is an open-label, single-arm study in patients with Idiopathic Pulmonary Fibrosis (IPF) aged 40 years and older.

The duration of study participation is approximately 20 weeks for each patient and comprises 6 study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult aged 40 years or older
2. Patient has signed written informed consent.
3. Patient has been diagnosed of IPF according to the most recent guideline on IPF diagnosis and management released by American Thoracic Society (ATS), European Respiratory Society (ERS), Japanese Respiratory Society (JRS), and Latin American Thoracic Association (ALAT).
4. Female patients of childbearing potential must have a negative urine pregnancy test and agree to use adequate birth control from screening throughout the study and for 30 days after the last study drug administration.
5. If a male patient has not been vasectomized at least 6 months before screening and partners with a woman of childbearing potential, he must be willing to use an acceptable contraceptive method throughout the study and for 30 days after the last study drug administration.

Exclusion Criteria:

1. Patient has a known diagnosis of a respiratory disorder other than IPF.
2. Substantial emphysema on high resolution computer tomography (HRCT) with degree of emphysema greater than fibrosis.
3. Patient is an active smoker.
4. Patient has evidence of active infection.
5. Patients currently has or has a history of cancer, except basal cell carcinoma or squamous cell carcinoma of the skin.
6. Patient has a concurrent medical or psychological condition that, in the investigator's opinion, may compromise the patient's ability to participate in the study or give informed consent, or may complicate the evaluations of the study drug.
7. Patient is receiving another investigational treatment for IPF at screening and/or plans to receive an investigational treatment for IPF during the current study.
8. Patient has chronic hepatitis or significantly elevated liver enzyme levels, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 × upper limit of normal (ULN) or total bilirubin above ULN.
9. Female patient who is pregnant, breast-feeding, or planning a pregnancy during the course of the study.
10. Woman of childbearing potential who is unwilling to use adequate birth control throughout the duration of the study.
11. Patient has participated in an investigational clinical trial during the last 4 weeks.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal laboratory values and/or adverse events that are related to treatment | 4 months

SECONDARY OUTCOMES:
Change from baseline on pulmonary function tests | 3 months
Change from baseline in imaging of thorax | 3 months
Change from baseline on biomarkers | 3 months

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec